CLINICAL TRIAL: NCT03126266
Title: ReRAD: A Phase II Canadian Pediatric Brain Tumour Consortium Study of Re-Irradiation as Treatment of Progressive or Recurrent Diffuse Intrinsic Pontine Glioma
Brief Title: Re-Irradiation of Progressive or Recurrent DIPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC16-0143
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Recurrent or Progressive Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Recurrence | interventions — Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving re-irradiation (Experimental): Patients will receive 30.6 Gy or 36 Gy of a second course of radiation therapy for progressive or recurrent DIPG
  Interventions: Radiation: re-irradiation

INTERVENTIONS:
Radiation: re-irradiation — if DIPG has progressed or recurred at 180 days or later from completion of primary radiation therapy, a second course of radiation therapy will be given

SUMMARY:
This is a single-arm, non-randomized study of re-irradiation of diffuse intrinsic pontine glioma (DIPG)

DETAILED DESCRIPTION:
Study therapy will consist of radiation therapy (RT) given over 17 treatment days (for 30.6 Gy in fractions of 1.8 Gy) or 20 treatment days (for 36 Gy in 1.8 Gy fractions), depending on the time from completion of the first course of RT. Treatment days will generally be weekdays, not including statutory holidays.

ELIGIBILITY:
Inclusion Criteria:

All of these criteria must be met for a patient to be eligible for this study:

1. Each site may accept a patient on study of any age that they have permission to treat and follow on study per their institutional policy.
2. The patient has no evidence of metastases on cranial or spinal MR imaging
3. The patient has received RT in the past, given to a total cumulative dose of <60 Gy; prior radiation using opposed lateral fields, conformal 3-D fields, IMRT or using protons is acceptable
4. At least 180 days have elapsed from the last day of primary RT for DIPG
5. The patient has recovered from all acute and subacute toxicities of prior RT and of chemotherapy, if chemotherapy was utilized in the past
6. The patient has been off all anti-tumour therapy for at least 14 days
7. The patient has a Lansky score of 40% or higher
8. The patient has a life expectancy anticipated to be at least 8 weeks with treatment using re-irradiation, with or without dexamethasone
9. The patient has no uncontrolled medical condition (e.g., seizures, diabetes, infection) that would interfere with the delivery of rRT
10. The patient agrees to not enroll on any other clinical trial of an anti-tumour intervention
11. The patient agrees to report and have recorded the use of all medications taken during ReRAD therapy, from the time of diagnosis of progression or recurrence, then through and after completion of, ReRAD therapy; this includes the use of complementary, alternative and dietary therapies
12. The patient is treated at a site where the study is approved by the local ethics board
13. Males and females of child-bearing potential must agree to use effective birth control measures during rRT
14. Consent, and, if applicable, assent, has been obtained according to institutional standards

Exclusion Criteria:

If the patient fulfills any of these criteria, then he or she will not be eligible for the study:

1. Females who are pregnant, due to risks from rRT on the developing fetus.
2. Any patient with a condition that prohibits the planned delivery of rRT as prescribed in this study.
3. Patients who are receiving any other clinical trial of an anti-tumour intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
second progression-free survival | up to 18 months from the start of re-irradiation
  length of time from start of re-irradiation to subsequent progression of disease

SECONDARY OUTCOMES:
overall survival | up to three years from initial diagnosis of DIPG
  time from initial diagnosis of DIPG to death following re-irradiation

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Lafay-Cousin, MD, Principal Investigator — University of Calgary
Locations (18):
- Australia (5):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Monash Children's Hospital, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital at London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU de Québec-Université Laval, Laval, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
- Starship Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No